CLINICAL TRIAL: NCT02894541
Title: A Randomized, Open-label, Single Dose, 1-sequence, 3-treatment, 3-period Crossover Study to Investigate the Effects of Food on the Pharmacokinetics/Pharmacodynamics of CKD-519 in Healthy Male Subjects
Brief Title: Study to Investigate the Effects of Food on the Pharmacokinetics/Pharmacodynamics of CKD-519
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 148FDI16004
Record Dates: First submitted 2016-09-05; First posted 2016-09-09 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2016-08

CONDITIONS: Healthy Volunteers
Keywords: Dyslipidemia; CKD-519; CETP inhibitor; Food Drug Interaction
MeSH Terms: conditions — Dyslipidemias | interventions — CKD-519

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- CKD-519 tablet 100mg (Experimental): CKD-519 tablet(formulation Ⅱ) 100mg(100mg X 1Tab) Period 1: CKD-519 100mg in fasted state Period 2:CKD-519 100mg with a standard meal Period 3:CKD-519 100mg with a high fat meal
  Interventions: Drug: CKD-519 100mg
- CKD-519 tablet 200mg (Experimental): CKD-519 tablet(formulation Ⅱ) 200mg(100mg X 2Tabs) Period 1:CKD-519 200mg in fasted state Period 2:CKD-519 200mg with a standard meal Period 3:CKD-519 200mg with a high fat meal
  Interventions: Drug: CKD-519 200mg
- CKD-519 soft capsule 100mg (Experimental): CKD-519 soft capsule(formulation Ⅲ) 100mg(100mg X 1Cap) Period 1:CKD-519 100mg in fasted state Period 2:CKD-519 100mg with a standard meal Period 3:CKD-519 100mg with a high fat meal
  Interventions: Drug: CKD-519 100mg
- CKD-519 soft capsule 200mg (Experimental): CKD-519 soft capsule(formulation Ⅲ) 200mg(100mg X 2Caps) Period 1:CKD-519 200mg in fasted state Period 2:CKD-519 200mg with a standard meal Period 3:CKD-519 200mg with a high fat meal
  Interventions: Drug: CKD-519 200mg

INTERVENTIONS:
Drug: CKD-519 100mg
  Other Names: CKD-519 tablet(formulation Ⅱ) 100mg(100mg X 1Tab)
  Arms: CKD-519 tablet 100mg
Drug: CKD-519 200mg
  Other Names: CKD-519 tablet(formulation Ⅱ) 200mg(100mg X 2Tabs)
  Arms: CKD-519 tablet 200mg
Drug: CKD-519 100mg
  Other Names: CKD-519 soft capsule(formulation Ⅲ) 100mg(100mg X 1Cap)
  Arms: CKD-519 soft capsule 100mg
Drug: CKD-519 200mg
  Other Names: CKD-519 soft capsule(formulation Ⅲ) 200mg(100mg X 2Caps)
  Arms: CKD-519 soft capsule 200mg

SUMMARY:
The purpose of this study is to investigate the effects of food on the pharmacokinetics/pharmacodynamics of CKD-519.

DETAILED DESCRIPTION:
A randomized, open-label, single dose, 1-sequence, 3-treatment, 3-period crossover study to investigate the effects of food on the pharmacokinetics/pharmacodynamics of CKD-519 in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

* Between 20 aged and 45 aged in healthy adult male
* Body weight more than 50, Body Mass Index between 18 and 29kg/m²
* Necessarily he agrees that use double contraceptions and do not sperm donation until two months during clinical trials and after the final dosage of investigational products
* Those who fully understand about this clinical trials after enough hearing, and then decided to join the clinical trials by themselves and to comply with the precautions written consent

Exclusion Criteria:

* Clinically significant disease with cardiovascular, respiratory, hepatobiliary, nephrological, hematological, gastrointestinal, endocrine, immune, integumentary, neurologic, psychiatric system
* Have a acute disease within 28 days before the beginning of study treatment
* Have a disease history that can effect drug absorption, distribution, metabolism, excretion
* Have a clinically significant chronic disease
* Systolic blood pressure<100mmHg or>140mmHg, diastolic blood pressure<60mmHg or>90mmHg
* Defined by the following 12-lead ECG, QTc>450msec
* Positive for serology test (HBsAg, anti-HCV Ab, anti-HIV Ab, VDRL(Venereal Disease Research Laboratories))
* Subject treated ethical drug within 14 days before the beginning of study treatment
* Subject treated over-the-counter or herbal medicine within 7 days before the beginning of study treatment
* Have a clinically significant allergic disease (except for mild allergic rhinitis, allergic dermatitis with no drugs)
* Cannot take standard Meal
* Whole blood donation within 60 days prior to the first dosing or component blood donation within 20 days prior to the first dosing
* Blood transfusion within 30 days
* Taking drugs have received any other investigational drug within 90 days prior to the first dosing
* Subject treated metabolizing enzyme inducers or inhibitors including barbiturates within 30 days
* Continuously taking caffeine(caffeine>5 cups/day), drinking alcohol(alcohol>210g/week), smoking excessive cigarettes(cigarette>10cigarettes/day)
* Impossible on who participants in clinical trial by investigator's decision including laboratory test result or another reasons(for example, noncompliance, a disobliging manner)

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Cmax of CKD-519 | 0(predose)~168
AUClast of CKD-519 | 0(predose)~168
Tmax of CKD-519 | 0(predose)~168
AUCinf of CKD-519 | 0(predose)~168
T1/2 of CKD-519 | 0(predose)~168
CL/F of CKD-519 | 0(predose)~168
Vd/F of CKD-519 | 0(predose)~168

SECONDARY OUTCOMES:
Inhibition of CETP(Cholesteryl ester transfer protein) Activity | 0(predose)~168

CONTACTS AND LOCATIONS:
Overall Officials: Ji Young Park, MD, PhD, Principal Investigator — Korea University
Locations (1):
- Korea university medical center, Seoul, Sungbuk-gu, South Korea

IPD SHARING:
Plan to Share IPD: No